CLINICAL TRIAL: NCT06645093
Title: Intermittent Fasting During Curatively Intended Chemotherapy for Malignant Lymphoma - a Randomized Feasibility Trial
Brief Title: Feasibility of Intermittent Fasting During Chemotherapy
Acronym: Fastestudien
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sonja H. Brunvoll, PhD, Postdoctoral researcher Sonja H. Brunvoll, PhD (co-PI together with Inger Ottestad, PhD), University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FasteStudien
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma; Cancer; Fasting
Keywords: Chemotherapeutic Toxicity; Chemotherapy; Adverse Effect; Short-term fasting; Feasibility studies; Fasting
MeSH Terms: conditions — Lymphoma; Neoplasms; Fasting; Intermittent Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Safety and feasibility study,-pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting group (Experimental): This group will fast 24 hours before and 24 hours after chemotherapy for all treatment cycles (4-6 cycles).
  Interventions: Other: Fasting
- Control group (No Intervention): This group will receive standard treatment, which include no fasting.

INTERVENTIONS:
Other: Fasting — Fasting implies 0 kilojoule. Water ad libitum is permitted.
  Arms: Fasting group

SUMMARY:
The goal of this randomized controlled parallel group trial is to examine if fasting before and after chemotherapy is safe, feasible and acceptable. The study population will include patients with either Hodgkin lymphoma or Diffuse Large B Cell Lymphoma.

The main questions aimed to answer are:

Whether fasting during chemotherapy is safe for patients, whether it is feasible to implement in a clinical setting, and whether patients find it acceptable.

We also want to examine a number of patient-reported outcome measures regarding health status and quality of life, such as dietary intake and adverse events from chemotherapy.

Researchers will compare fasting to standard treatment.

Participants will:

* Fast 24 hours before and 24 hours after chemotherapy in addition to standard treatment or receive only standard treatment
* Keep a diary of their dietary intake 24 hours before and 24 hours after chemotherapy
* Keep a diary of their dietary intake for three consecutive days between chemotherapy cycles
* Answer questionnaires/questions in relation to side effects from fasting, side effects/adverse events of chemotherapy, quality of life
* Take bioimpedance analysis (including body mass index and body composition)
* Take blood- and feces samples

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diffuse large B-cell lymphoma planned to receive R-CHOP (rituximab, vincristine, doxorubicin, cyclophosphamide, and prednisolone) and Hodgkin lymphoma receiving ABVD (doxorubicin, bleomycin, vinblastine and dacarbazine)
* Age ≥ 18 years
* ECOG status 0-2
* Normal weight and overweight (BMI ≥ 18,5 kg/m^2)

Exclusion Criteria:

* Receiving concurrent radiation therapy and/or treatment
* Other concomitant disease that may make intermittent fasting complicated such as diabetes mellitus
* ECOG status: > 3
* BMI < 18,5 kg/m2
* Age > 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety, measured as 1) number of adverse events | 1 year
  To test whether fasting is safe. 1) Explored by investigating adverse events from intermittent water-only fasting
Safety, measured as 2) changes in body weight | 1 year
  To test whether fasting is safe. 2) by investigating changes in body weight throughout the treatment comparing the intervention and control groups.
Feasibility,- measured by 1) recruitment (attrition rate) | 1 year
  Whether fasting is feasible. Explored in order to determine whether a larger trial can be successfully conducted in a similar setting with lymphoma patients fasting during cancer treatment.
Feasibility,- measured as 2) compliance | 1 year
  Whether fasting is feasible. Explored in order to determine whether a larger trial can be successfully conducted in a similar setting with lymphoma patients fasting during cancer treatment.
Acceptability,- patient burden, acceptance and experience | 1 year
  Whether fasting is acceptable. Explored from a perspective of the participant, as the degree to which patients find the trial, its procedures, and its interventions agreeable, suitable, and satisfactory during chemotherapy treatment

SECONDARY OUTCOMES:
Adverse events from chemotherapy | 1 year
  Adverse events including number of infections, graded according to Common Terminology Criteria for Adverse Events
Toxicity, including hematological toxicity and standard organ toxicity | 1 year
  Evaluation of toxicity, including hematological toxicity and other relevant organ toxicities with blood test and using computer tomography (CT) or fluoro-deoxy-glucose positron emission tomography computer tomography (FDG-PET-CT)
Health-Related Quality of Life | 1 year
  By using EORTC QLQ-C30 questionnaire
Nutritional impact symptoms | 1 year
  The linguistic and content validation of the translated and culturally adapted Patient Generated Subjective Global Assessment (PG-SGA) will be utilized for gathering data on nutritional impact symptoms
Dietary intake | 1 year
  Dietary intake 24 hours before and 24 hours after chemotherapy and the usual intake between chemotherapy cycles using food diary.
Weight loss, body mass index (BMI) and body compositon | 1 year
  Bioelectrical impedance (BIA) will be used to collect data to explore changes in body weight, BMI and body composition.
Unplanned readmissions and hospitalization | 1 year
  In terms of numbers of readmissions, unplanned out- or inpatient visits, and days in the hospital

OTHER OUTCOMES:
Mechanistic aspects of fasting | 1 year
  To better understand nutrition and metabolism related to fasting and cancer, we want to examine various biomarkers related to glucose, amino acid and fat metabolism, and inflammation, such as e.g. glucose, insulin, amino acids, triglycerides, C-reactive protein (CRP).
Fasting and microbiota | 1 year
  We will analyze the gut microbiota to explore the effect of fasting on the gut microbiota. We will collect feces samples at start and end of treatment to characterize the microbiota using high throughput sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Brunvoll, PhD, Principal Investigator — Department of Nutrition, University of Oslo; Inger Ottestad, PhD, Principal Investigator — Department of Nutrition, University of Oslo
Locations (1):
- Department of Nutrition, University of Oslo, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No